CLINICAL TRIAL: NCT05118022
Title: Artificial Intelligence Identified Dyskalemia Using Electrocardiogram (AIDE) Prompts Immediate Treatment
Brief Title: Artificial Intelligence Identified Dyskalemia Using Electrocardiogram (AIDE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NDMC2021004
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hyperkalemia; Hypokalemia
MeSH Terms: conditions — Hyperkalemia; Hypokalemia | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to intervention will be cared by physicians under AI-ECG support.
  Interventions: Other: Artificial Intelligence identified Dyskalemia using Electrocardiogram (AIDE) system
- Control (No Intervention): Patients randomized to control will be cared by routine practice.

INTERVENTIONS:
Other: Artificial Intelligence identified Dyskalemia using Electrocardiogram (AIDE) system — Once the AIDE indicates high risk of dyskalemia, an obvious message by scarlet letter was appeared in the HIS operation interface to corresponding physicians. To avoid the alert fatigue, we selected the cut-off points with expected positive predictive values of ≥40% according to previous data, which was the consensus of enrolled physicians before the trial considering the clinical loading. The physicians received the AIDE alerts as long as they were operating HIS logged in by their account, even if they were caring other patients. Physicians can review the AIDE predictions of patients in the intervention group. Therefore, this was a single-blind study since HIS presented different information for patients in intervention and control groups. The participated physicians understood the likelihood of dyskalemia and cardiac risk for those patients with ECG-dyskalemia, and provided suitable medical care according to patients' conditions.
  Arms: Intervention

SUMMARY:
This is a randomized controlled trial (RCT) to test a novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool for improving the diagnosis and management of potassium abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients in emergency department.
* Patients recieved at least 1 ECG examination.

Exclusion Criteria:

* Patients recieved dyskalemia-related treatment before ECG examination.
* The patients recieved ECG at the period of inactive AI-ECG system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14989 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Cumulative proportion of hyperkalemia treatment | Within 3 hours
  Calcium supplement, insulin, potassium binding resin, β2-agonist, loop diuretics, sodium bicarbonate, and hemodialysis.
Cumulative proportion of hypokalemia treatment | Within 3 hours
  Intravenous potassium chloride, oral potassium gluconate, and oral potassium chloride

SECONDARY OUTCOMES:
Cardiac arrest (sudden death) | Within 3 days
  Cardiac arrest (sudden death)
Cumulative proportion of All-cause mortality | Within 365 days
  All-cause mortality
Cumulative proportion of electric shock | Within 6 hours
  Cardioversion
Cumulative proportion of CPR event | Within 6 hours
  Cardiopulmonary pesuscitation
Cumulative proportion of Discharge | Within 14 days
  Discharge from inpatient department or emergency department
Cumulative proportion of Treatment-induced hypokalemia event | Within 24 hours
  Treatment-induced hypokalemia event
Cumulative proportion of Treatment-induced hyperkalemia event | Within 24 hours
  Treatment-induced hyperkalemia event

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin C, Lin CS, Chen SJ, Tsai SH, Sung CC, Chen CC, Hsu YJ, Hung YJ, Lin SH. AI-enabled electrocardiogram alert for potassium imbalance treatment: a pragmatic randomized controlled trial. Nat Commun. 2026 Jan 8;17(1):159. doi: 10.1038/s41467-025-66394-4. PMID 41507124